CLINICAL TRIAL: NCT04419805
Title: Single Palatal Temporary Anchorage Device for Anterior Open Bite: a Randomized Clinical Trial
Brief Title: Single Palatal Temporary Anchorage Device for Anterior Open Bite
Acronym: SPaTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Peter Mossey, Professor, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-054-19
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Anterior Openbite
Keywords: Orthodontics; Temporary Anchorage Device; Anterior Open Bite

STUDY DESIGN:
Intervention Model Description: Randomised parallel 2 group clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blind to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Palatal TAD (Experimental): Single Palatal TAD for orthodontic molar intrusion
  Interventions: Device: Single Palatal TAD
- Two buccal TADs (Experimental): Two buccal TADs for orthodontic molar intrusion
  Interventions: Device: Two buccal TADs

INTERVENTIONS:
Device: Single Palatal TAD — A single mini-screw inserted in the mid-palate
  Arms: Single Palatal TAD
Device: Two buccal TADs — Two buccal TADs inserted in the upper jaw
  Arms: Two buccal TADs

SUMMARY:
Participants are orthodontic patients with anterior open bite (AOB) malocclusion. These patients will be treated by molar intrusion achieved using one of two interventions, either orthodontic fixed appliances incorporating a single palatal Temporary Anchorage Device (TAD) or orthodontic fixed appliances incorporating two buccal TADs

DETAILED DESCRIPTION:
Participants will be recruited from those attending Dundee Dental Hospital Orthodontic Department and those currently awaiting treatment. Those that meet the inclusion and exclusion criteria will be invited to participate. After obtaining consent they will be allocated to receive one of the two interventions. The two interventions represent the currently available options for treatment of mild - moderate (1-6mm) anterior open bite in the Orthodontic Department and as such patients will be receiving routine treatment regardless of the arm they are randomised to. In order to assess the more effective intervention additional records will be taken during the treatment involving additional cephalometric radiographs, additional intra-oral scans or dental impressions (See later for details). Primary outcome is at the end of intrusion with TADs after 9-12 months, but participants will be followed until completion of treatment for the secondary outcome of stability of intrusion and overbite correction

ELIGIBILITY:
Inclusion Criteria:

* Patients with AOB of 1-6mm
* Aged between (12 and 40 years).
* Able to consent.
* Patient due to undergo orthodontic treatment with fixed orthodontic braces.

Exclusion Criteria:

* Patient has previously had upper first permanent molar extraction.
* Patient with congenital cleft of lip and/or palate or any other craniofacial anomalies.
* Patient with bone disease or taking medications that affect the bone quality or nature.
* Patient with an active digit sucking habit.
* Pregnant or breastfeeding women

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Molar intrusion | 9-12 months after treatment commences
  Amount of upper molar intrusion measured in mms on cephalometric radiograph

SECONDARY OUTCOMES:
Overbite (vertical overlap of anterior teeth) | 9-12 months after treatment commences
  Change in overbite (vertical overlap of anterior teeth) measured clinically directly from the teeth with a ruler and on 3D dental scans using 3D analysis software, both in mms
Patient Experience | 9-12 months after treatment commences
  Patient experience with the use of temporary anchorage devices for intrusion by validated questionnaire which uses 3 or 4 point Likert Scales for a range of questions across relevant doamins. Depending on the question the scales are 'Improved/Same/Worse/Much worse' or 'Not at all / A little / A lot' or 'I do more / no difference / I do less' (Yassir et al 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mossey, BDS, Principal Investigator — University of Dundee
Locations (1):
- Dundee Dental Hospital, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yassir YA, McIntyre GT, Bearn DR. Three questionnaires to assess the perception of fixed orthodontic therapy before, during and after treatment: validity and reliability. Eur J Orthod. 2017 Aug 1;39(4):402-410. doi: 10.1093/ejo/cjw076. PMID 27864320